CLINICAL TRIAL: NCT02444442
Title: The Australian SHAM Controlled Clinical Trial of Renal DeNervation in Patients With Resistant Hypertension (AUSHAM-RDN-01)
Brief Title: Sham Controlled Clinical Trial of Renal Denervation in Patients With Resistant Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002/15
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
Keywords: Renal denervation; Blood pressure; Cardiovascular risk; Target organ damage; Sympathetic activity; Non-compliance
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal Denervation (Active Comparator): participants randomised to undergo renal denervation
  Interventions: Device: Renal Denervation
- Sham control (Sham Comparator): participants randomised to undergo sham procedure
  Interventions: Other: Sham control

INTERVENTIONS:
Device: Renal Denervation — Deliberate disruption of the renal nerves via radio frequency energy delivery to renal arteries.
  Arms: Renal Denervation
Other: Sham control — Arterial access only. No delivery of radio frequency energy to renal arteries.
  Arms: Sham control

SUMMARY:
The purpose of this study is to assess the efficacy of catheter-based renal denervation in reducing blood pressure in patients with resistant hypertension compared to a sham procedure. Patients will be randomized to RDN or sham control in a 2:1 ratio. All participants will be switched to a single pill triple combination treatment prior to the procedure.

A total of 105 patients will be recruited into the study, 70 patients in the RDN arm and 35 patients in the sham control arm.

The duration of this study is 36 months.

ELIGIBILITY:
Inclusion Criteria:

* systolic office BP ≥140mmHg and ambulatory day time average ≥135mmHg despite concurrent treatment with ≥3 anti-hypertensive drugs

Exclusion Criteria:

* renal artery anatomy ineligible for treatment
* eGFR <15mL/min/1.73m2 (using MDRD calculation)
* myocardial infarction, unstable angina or cerebrovascular accident within 3 months of screening visit
* life expectancy of <12 months
* female participants of childbearing potential must have negative pregnancy test prior to treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Change in ambulatory systolic blood pressure between groups | 6 months post procedure
  Difference in mean ambulatory systolic daytime blood pressure between RDN group and sham-control group at 6 month follow up.

SECONDARY OUTCOMES:
Change in mean 24h systolic blood pressure between groups | 6 months post procedure
  Change in mean 24h systolic blood pressure between RDN group and sham-control group at 6 month follow up.
Change in mean night time systolic blood pressure between groups | 6 months post procedure
  Change in mean night time systolic blood pressure between RDN group and sham-control group at 6 month follow up.
Change in mean office systolic blood pressure between groups | 6 months post procedure
  Change in mean office systolic blood pressure between RDN group and sham-control group at 6 month follow up.

OTHER OUTCOMES:
Change in percentage of patients achieving BP target between groups | 6 months post procedure
  Change in percentage of patients achieving BP target between groups
Change in percentage of patients with an ambulatory systolic BP reduction ≥5mmHg between groups | 6 months post procedure
  Change in percentage of patients with an ambulatory systolic BP reduction ≥5mmHg between groups
Change in percentage of patients with an office systolic BP reduction ≥10mmHg between groups | 6 months post procedure
  Change in percentage of patients with an office systolic BP reduction ≥10mmHg between groups
Change of sympathetic nerve activity between groups | 6 months post procedure
  Change of sympathetic nerve activity (MSNA, renal and whole body NE spillover) between groups
Change in left ventricular function between groups | 6 months post procedure
  Change in left ventricular function (LV mass index, ejection fraction, diastolic filling) between groups
Change in Serum Biochemistry between groups | 6 months post procedure
  Plasma Renin Activity, aldosterone levels, estimated Glomerular Filtration Rate(eGFR), inflammatory markers, fasting glucose, fasting insulin, C-peptide, Homeostasis Model Assessment (HOMA) index, Lipid profile between groups
Change in Urine Biochemistry between groups | 6 months post procedure
  Urinary albumin creatinine ratio (UACR), 24 hour urinary creatinine clearance, sodium between groups
Change in Quality of Life between groups | 6 months post procedure
  Change in Quality of life as assessed by relevant questionnaires between groups
Change in cognitive function between groups | 6 months post procedure
  Change in cognitive function as assessed by relevant questionnaires and assessment tools between groups
Change in microRNA expression between groups | 6 months post procedure
  Change in microRNA expression as assessed by relevant assays between groups

CONTACTS AND LOCATIONS:
Overall Officials: Markus P Schlaich, Professor, Principal Investigator — Laboratory Head, Neurovascular Hypertension and Kidney Disease (Baker IDI)
Locations (1):
- Baker IDI Heart & Diabetes Institute, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Pisano A, Iannone LF, Leo A, Russo E, Coppolino G, Bolignano D. Renal denervation for resistant hypertension. Cochrane Database Syst Rev. 2021 Nov 22;11(11):CD011499. doi: 10.1002/14651858.CD011499.pub3. PMID 34806762